CLINICAL TRIAL: NCT01578187
Title: Evaluating Label Comprehension and Usability of the Hair2Go System
Brief Title: Hair2Go Label Comprehension and Usability Study
Acronym: OHR6-LCU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: OHR6-LCU
Record Dates: First submitted 2012-04-13; First posted 2012-04-16 (Estimated); Results first posted 2013-10-11 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-11

CONDITIONS: Hair Removal
Keywords: hair reduction; hair removal; hair clearance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hair2Go device (Experimental)
  Interventions: Device: Hair2Go

INTERVENTIONS:
Device: Hair2Go — Treatment with the device once under observation
  Other Names: Mē my elōs

SUMMARY:
The purpose of this study is to test label comprehension and usability of the hair removal device in 60 male and female participants. The study population will represent the US demographic distribution of skin types and will include varying levels of literacy.

DETAILED DESCRIPTION:
This will be a single-visit study consisting of two phases: Phase I - assessing label comprehension and Phase II - usability. For Phase I, subjects will be asked to review the outer packaging of the mē device. Each subject will be taken through an interview which will evaluate messages on the external product labeling regarding product use and self-selection criteria. Subjects, who are not self-excluders and/or contraindicated for use of the device will continue with Phase II of the study. This usability phase will consist of watching the instructional DVD, reading the User Guide and then performing a skin sensitivity test. Subjects will be expected to self-administer the hair removal treatment in a simulated home-use environment under observation of the study personnel. The users will have a telephone in the room and may call a phone number and request assistance while performing the treatment, simulating the toll-free hotline that will be available to consumers in commercial use.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, between 18 and 65 years of age.
2. Able to read and understand the written consent form.
3. Willing to sign informed consent.
4. Able to read and speak English.
5. Willing and able to participate in the study procedures.

Exclusion Criteria:

1. The participant or anyone in their household is currently employed by a marketing research department or company, an advertising agency or public relations firm, a pharmaceutical company, a healthcare device manufacturer, a cosmetic or personal care company.
2. The participant is currently employed at a salon, day spa or beauty school/college as a stylist, barber, esthetician or beauty instructor.
3. The respondent has ever been trained or employed as a healthcare professional.
4. The participant normally wears corrective lenses, contacts or glasses to read and does not bring them with him/her to the study site.
5. The participant has participated in any market research study, product label study or clinical trial in the past thirty (30) days.
6. Non-English speakers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2012-03; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Caswell, Ph.D., Principal Investigator — Consumer Product Testing Company
Locations (1):
- Consumer Product Testing Company, Fairfield, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at a single site specialized in consumer product testing.
Groups:
- Hair2Go Device: This group included subjects who participated in the label comprehension phase. From these subjects, 48 subjects self-included in the usability phase (no contraindications) and chose to use the device for 1 treatment.
  The subjects included all skin types and a population of low health literacy subjects based on the Rapid Estimate of Adult Literacy in Medicine (REALM) test.
Period: Label Comprehension Phase
Arm/Group | Hair2Go Device
Started | 63
Completed | 63
Not Completed | 0
Period: Usability Phase
Arm/Group | Hair2Go Device
Started | 48
Completed | 47
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Hair2Go Device: The subjects who participated in the label comprehension phase, of them most participated in the usability phase. The subjects included all skin types and a population of low health literacy subjects based on the Rapid Estimate of Adult Literacy in Medicine (REALM)test.
Arm/Group | Hair2Go Device
Number analyzed (Participants) | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 63
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 63

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Correctly Determining Eligibility for Use of the Device (Responders)
Description: Label comprehension will be based on responses to a questionnaire. Questions will be based on a tiered system by level of importance in responding correctly according to the following:
  1. Questions regarding safe use of the system.
  2. Questions regarding correct use of the system(not related to safety).
  In order to demonstrate how well the label instruction, as a whole, was understood by all subjects, the proportion of subjects who correctly understood the label as a whole was calculated by classifying each subject as either a "responder" or "non-responder" based on the following criteria regarding all questions:
  A subject was considered a responder if he/she correctly answered 11/12 questions related to safety AND 5/6 low category questions not related to safety.
  The study was considered a success if the response rate (i.e., the proportion of subjects correctly understanding the label based on the responder criteria) was at least 90%.
Time Frame: 1 hour
Population: Sample size was discussed with the FDA during a pre-IDE teleconference
Measure: Number; unit: percentage of participants
Groups:
- Label Comprehension Group: Subjects that participated in the label comprehension phase of the study
Arm/Group | Label Comprehension Group
Number analyzed (Participants) | 63
percentage of participants | 94

2. Primary Outcome: Percentage of Participants Performing Critical/Non-critical Errors
Description: Study staff will record the number of errors according to the following:
  1. Critical error: an error that may cause a serious adverse event or an adverse event from a single occurrence
  2. Non critical error: An error that, if repeated without correction/intervention, may cause an adverse event.
Time Frame: 1-2 hours
Population: Subjects who were not self-excluders in the label comprehension phase and consented to continue to the usability phase (product use).
Measure: Number; unit: percentage of participants with errors
Groups:
- Usability - Critical Error: Critical error: an error that may cause a serious adverse event or an adverse event from a single occurrence
- Usability - Non Critical Error: Non critical error: An error that, if repeated without correction/intervention, may cause an adverse event.
Arm/Group | Usability - Critical Error | Usability - Non Critical Error
Number analyzed (Participants) | 47 | 47
percentage of participants with errors | 0 | 2.1

ADVERSE EVENTS:
Time Frame: This was a single visit study
Description: The label comprehension phase of the study did not involve a treatment with the device. Of the 63 participant of the label comprehension phase, 47 subjects who were not self-excluders continued to the usability phase that included a treatment. Therefore the number of "at risk" individuals is 47 and not the original 63.
Groups:
- Hair2Go (Me) Device: The subjects who participated in the label comprehension phase; the majority of whom participated in the usability phase. The subjects included all skin types and a population of low health literacy subjects based on the Rapid Estimate of Adult Literacy in Medicine (REALM)test.
Arm/Group | Hair2Go (Me) Device
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No